CLINICAL TRIAL: NCT04184232
Title: Treatment of Recurrent Bladder Cancer With Autologous Monocyte-derived Dendritic Cells
Brief Title: Treatment of Recurrent Bladder Cancer With Dendritic Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_DC1(BLAD)
Record Dates: First submitted 2019-12-01; First posted 2019-12-03 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Dendritic cells
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dendritic cells (Experimental): Patients with the recurrent bladder cancer receiving standard treatment and autologous dendritic cells
  Interventions: Biological: Dendritic cells; Other: Standard treatment according to the Clinical protocols
- Control (Active Comparator): Patients with the recurrent bladder cancer receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Dendritic cells — Autologous dendritic cells primed with muc-1/wt-1 peptides
  Arms: Dendritic cells
Other: Standard treatment according to the Clinical protocols — Standard treatment of bladder cancer according to the Clinical protocols

SUMMARY:
Treatment of recurrent bladder cancer with dendritic cells

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of pTa bladder cancer;
* Patient who require repetitive transurethral resection;
* Expression of muc-1/wt-1 by the tumor;
* EGOC 0-3;

Exclusion Criteria:

* any medical condition which can be associated with the high risk for the patient;
* pregnancy/lactation;
* chronic infections, including hepatitis B/C, tuberculosis, HIV

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation | 1 year
  1 year relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — Director, the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Alexander V Prokharau, Dr, Study Director — Head of the chair, Belarusian State Medical University
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No